CLINICAL TRIAL: NCT03008317
Title: Microbial Adhesion to Metallic Versus Non Metallic Surfaces of Bounded Removable Partial Denture
Acronym: splitmouth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hager essam el azizi, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBC-CU-2016-12-164
Record Dates: First submitted 2016-12-20; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Polyetheretherketone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- non metallic (Active Comparator): PEEK denture base,
  Interventions: Device: PEEK
- metallic denture base (Placebo Comparator): cobalt chromium alloy denture base
  Interventions: Device: PEEK

INTERVENTIONS:
Device: PEEK — a metallic denture base
  Other Names: polyetheretherketone denture base; cobalt chromium alloy denture base

SUMMARY:
a split mouth randomized clinical trial that compares quantity and quality of bacterial adhesion under both PEEK versus cobalt chromium alloy denture base.

DETAILED DESCRIPTION:
this study aimed to compare the adhesion of microorganisms to the non metallic denture base of PEEK and metallic denture base of cobalt chromium alloy in patients with class III modification 1

ELIGIBILITY:
Inclusion Criteria:

* patients are medically free

Exclusion Criteria:

* patients with badly broken abutments

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
microbial culture using number of clonies after insertion by 3 months | one year
  microbial adhesion will be measured using continous cultures to assess number of colonies

IPD SHARING:
Plan to Share IPD: Undecided